CLINICAL TRIAL: NCT06192316
Title: Human Laboratory Study of the Effects of Nicotine Product Claims on Appeal, Perceptions, and Use Behavior
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Darren Mays, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OSU-23115; NCI-2023-08947 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); U54CA287392 (NIH)
Record Dates: First submitted 2023-12-13; First posted 2024-01-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Behavior, Risk
Keywords: oral nicotine pouch; cancer control; cancer prevention
MeSH Terms: conditions — Risk-Taking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (9):
- Nicotine Concentration: None Displayed; Nicotine Source Claim 1 (Experimental): Participants view randomized images of nicotine-containing product packaging and complete a lapse task test on study. Participants also complete questionnaires on study.
  Interventions: Behavioral: 3x3 between-subjects experimental exposure
- Nicotine Concentration: None Displayed; Nicotine Source Claim 2 (Experimental): Participants view randomized images of nicotine-containing product packaging and complete a lapse task test on study. Participants also complete questionnaires on study.
  Interventions: Behavioral: 3x3 between-subjects experimental exposure
- Nicotine Concentration: None Displayed; Nicotine Source Claim 3 (Experimental): Participants view randomized images of nicotine-containing product packaging and complete a lapse task test on study. Participants also complete questionnaires on study.
  Interventions: Behavioral: 3x3 between-subjects experimental exposure
- Nicotine Concentration: Low; Nicotine Source Claim 1 (Experimental): Participants view randomized images of nicotine-containing product packaging and complete a lapse task test on study. Participants also complete questionnaires on study.
  Interventions: Behavioral: 3x3 between-subjects experimental exposure
- Nicotine Concentration: Low; Nicotine Source Claim 2 (Experimental): Participants view randomized images of nicotine-containing product packaging and complete a lapse task test on study. Participants also complete questionnaires on study.
  Interventions: Behavioral: 3x3 between-subjects experimental exposure
- Nicotine Concentration: Low; Nicotine Source Claim 3 (Experimental): Participants view randomized images of nicotine-containing product packaging and complete a lapse task test on study. Participants also complete questionnaires on study.
  Interventions: Behavioral: 3x3 between-subjects experimental exposure
- Nicotine Concentration: High; Nicotine Source Claim 1 (Experimental): Participants view randomized images of nicotine-containing product packaging and complete a lapse task test on study. Participants also complete questionnaires on study.
  Interventions: Behavioral: 3x3 between-subjects experimental exposure
- Nicotine Concentration: High; Nicotine Source Claim 2 (Experimental): Participants view randomized images of nicotine-containing product packaging and complete a lapse task test on study. Participants also complete questionnaires on study.
  Interventions: Behavioral: 3x3 between-subjects experimental exposure
- Nicotine Concentration: High; Nicotine Source Claim 3 (Experimental): Participants view randomized images of nicotine-containing product packaging and complete a lapse task test on study. Participants also complete questionnaires on study.
  Interventions: Behavioral: 3x3 between-subjects experimental exposure

INTERVENTIONS:
Behavioral: 3x3 between-subjects experimental exposure — Participants will be randomly assigned to conditions in a 3 (Nicotine Concentration: None on label, Low, High) x 3 (Nicotine Source Claim: None, "Tobacco Free," "Synthetic Nicotine") between-subjects design. We will stratify randomization by young adult susceptible non-users and adult tobacco users for balance across the conditions. Participants will view 16 oral nicotine pouch pack images in random order that correspond to the nicotine concentration and source claim condition they are randomized to. Within each condition, pack images will vary by 4 brands and 4 flavors per brand. While viewing the images, we will collect psychophysiological data including heart rate, galvanic skin response, and eye tracking.

SUMMARY:
This study evaluates knowledge, feelings and thoughts regarding nicotine products among young adults who are susceptible to but do not use tobacco/nicotine and adults who use tobacco/nicotine.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Examine the effects of nicotine concentration and source claims on engagement with ONP packaging using laboratory-based psychophysiological assessment.

II. Examine the effects of nicotine concentration and source claims on participant self-reported ONP perceptions, behavioral intentions, and ONP trial.

This is an experimental behavioral study. Participants view randomized images of nicotine-containing product packaging and complete a lapse task test on study. Participants also complete questionnaires on study.

ELIGIBILITY:
Inclusion Criteria:

* Young adult susceptible non-users aged 18-24 who have never used ONPs and have never used but are susceptible to using either:

  * combustible tobacco only (cigarettes, cigars, waterpipe)
  * non-combustible tobacco only (ST, ECs, heated tobacco products)
  * or both combustible and non-combustible tobacco (i.e., dual susceptibility)
* Adult tobacco users aged 18-65 who have never used ONPs OR have used ONPs >3 months ago and 10 times or less in their lifetime. All adult tobacco users must also be:

  * exclusive combustible tobacco users
  * exclusive non-combustible tobacco users
  * dual users

    * For adult tobacco users, we will define current use as use of combustible and/or non-combustible tobacco every day or some days for 6 months or longer
* Willing and able to complete an in-person lab visit.

Exclusion Criteria:

* Age < 18 or > 65
* Are not susceptible non-users or current tobacco users
* Are unwilling or unable to complete and in person lab visit.
* Have used ONPs within the past 3 months
* Have used ONPs more than 10 times in their lifetime

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2028-09-14 (Estimated); Study Completion 2028-09-14 (Estimated)

PRIMARY OUTCOMES:
Visual Attention - Dwell Time | 1 day (Single Time Point: During Exposure)
  Visual attention will be measured via eye movements using SmartEye AI-X eye tracker with a 60 Hz sampling rate. Areas of interest (AOIs) will be predefined for each pack image including: 1) Full pack image; 2) Nicotine concentration; 3) Nicotine source claim; 4) Branding (i.e., brand name, flavors); 5) Warning label. A primary outcome for visual attention will be dwell time on AOIs.
Visual Attention - Time to First Fixation | 1 day (Single Time Point: During Exposure)
  Visual attention will be measured via eye movements using SmartEye AI-X eye tracker with a 60 Hz sampling rate. Areas of interest (AOIs) will be predefined for each pack image including: 1) Full pack image; 2) Nicotine concentration; 3) Nicotine source claim; 4) Branding (i.e., brand name, flavors); 5) Warning label. A primary outcome for visual attention will be time to first fixation on AOIs.
Visual Attention - Number of Fixations | 1 day (Single Time Point: During Exposure)
  Visual attention will be measured via eye movements using SmartEye AI-X eye tracker with a 60 Hz sampling rate. Areas of interest (AOIs) will be predefined for each pack image including: 1) Full pack image; 2) Nicotine concentration; 3) Nicotine source claim; 4) Branding (i.e., brand name, flavors); 5) Warning label. A primary outcome for visual attention will be number of fixations (i.e., saccades) to AOIs.
Cognitive Attention | 1 day (Single Time Point: During Exposure)
  Conceptualized as the cognitive resources allocated to encode a message into working memory, attention will be operationalized as the difference in heart rate (HR) between a baseline period prior to each pack image and during each second of the pack image exposure assessed with ECG. Beats per minute (BPM) will be collected with the Shimmer3 sampled at 512 Hz. This is an established psychophysiological measure of cognitive resources devoted to stimuli processing.
Arousal | 1 day (Single Time Point: During Exposure)
  Arousal is an indicator of physiological activation of the sympathetic nervous system and will be measured by skin conductance using Shimmer3 Galvanic Skin Response EDA sensors sampled at 128 Hz
Recall | 1 day (Single Time Point: During Exposure)
  We will capture unaided recall, a measure of storage in memory, via 3 open ended questions on a questionnaire pertaining to nicotine concentration, brand names, and source information corresponding to conditions to which participants are randomized. Responses will be coded, and coding reliability will be established, to create a score with higher values reflecting better recall of information about nicotine dimensions in the stimuli.
ONP Perceptions | 1 day (Single Time Point: During Exposure)
  We will capture perceptions of ONPs with 7 items that align with expert recommendations for assessing cognitive and affective aspects of tobacco risk perceptions. Items will assess perceived risk of health harm from ONPs, perceived risk of addiction from ONPs, worry about harm, and worry about addiction. The items are on a 1-7 response scale, have excellent reliability, and are averaged to create an overall score.
ONP Perceptions Relative to Other Products | 1 day (Single Time Point: During Exposure)
  We will also capture perceived harm and addictiveness of ONPs relative to cigarettes, smokeless tobacco, and electronic cigarettes using valid items on a 1-5 response scale.
ONP Intentions | 1 day (Single Time Point: During Exposure)
  We will assess curiosity, interest, and likelihood of using ONPs post-exposure. These are valid predictors of future use of novel tobacco and nicotine products among never users. Items are on a 1-7 scale, have excellent reliability, and are combined to create an overall ONP intentions score.

OTHER OUTCOMES:
ONP Trial (Lapse Task) | Single Time Point for 25 Minutes
  This is a valid behavioral measure that was originally developed for smoking cue reactivity research and used in prior work by others and our team. The lapse task will assess ONP trial, time to trial, and ONP product selection.

CONTACTS AND LOCATIONS:
Overall Officials: Darren Mays, MPH, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
We will consider requests to share de-identified individual participant data by request and according to the investigator's study protocol and institutional data sharing policy.

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu